CLINICAL TRIAL: NCT07089186
Title: A Phase 3, Multicenter, Randomized, Open-label, Active-controlled, Parallel-design Clinical Study to Evaluate the Efficacy and Safety of Meropenem and Pralubactam for Injection in the Treatment of Carbapenem-Resistant Enterobacteriaceae Infections
Brief Title: Study to Assess the Efficacy and Safety of Meropenem and Pralurbactam in Carbapenem-Resistant Enterobacteriaceae Infections
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FL058-302
Record Dates: First submitted 2025-06-25; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Hospital-acquired Bacterial Pneumonia (HABP); Ventilator-associated Bacterial Pneumonia (VABP); Complicated Intra-abdominal Infection (cIAI); Complicated Urinary Tract Infection (cUTI); Bloodstream Infection (BSI)
MeSH Terms: conditions — Sepsis | interventions — Meropenem; Colistin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem and Pralurbactam (Experimental): Meropenem and Pralurbactam (180min infusion)
  Interventions: Drug: Meropenem and Pralurbactam
- Best Available Therapy (Active Comparator): Subjects will receive Best Available Therapy (IV antibiotics)
  Interventions: Drug: Best Available Therapy (e.g., colistin, meropenem, tegecycline, amikacinceftezidime-avibatam)

INTERVENTIONS:
Drug: Meropenem and Pralurbactam — 3g，q8h，180min infusion，Dose adjustments are available for participants with eGFR(mL/min)
  Arms: Meropenem and Pralurbactam
Drug: Best Available Therapy (e.g., colistin, meropenem, tegecycline, amikacinceftezidime-avibatam) — The main therapeutic agents anticipated for use, either in combination or as monotherapy, commonly include colistin, meropenem, tigecycline, amikacin, and ceftazidime-avibactam.
  Arms: Best Available Therapy

SUMMARY:
The study will evaluate the efficacy and safety of Meropenem and Pralurbactam versus Best Available Therapy in the treatment of Carbapenem-Resistant Enterobacteriaceae Infections. Infections evaluated in the study will be hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), complicated intra-abdominal infection (cIAI), complicated urinary tract infection (cUTI), and Bloodstream Infection (BSI).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female≥18 and ≤80 years of age，
* Participant must have a diagnosis of an infection (HABP/VABP, cUTI, cIAI, BSI) due to confirmed Carbapenem-Resistant Enterobacteriaceae infection, requiring administration of IV antibacterial therapy
* Participant who had received appropriate prior empiric antibacterial therapy for a carbapenem-resistant pathogen must meet at least 1 of the following criteria: no or no more than 24h; worsening of objective symptoms or signs after at least 48 hours of antibacterial therapy; no change of objective symptoms or signs after at least 72 hours of antibacterial therapy
* The estimated survival time is more than 28 days
* Understand and abide by the research procedures and methods, voluntarily participate in this research, and sign an informed consent form

Exclusion Criteria:

* Participants who need more than 3 systemic antibiotics as part of best available treatment (BAT)
* Participant is expected to require more than 21 days of treatment
* Acute Physiology and Chronic Health Evaluation (APACHE) II score >30 using the most recent available data
* Other medical or psychiatric condition may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Those who participated in other clinical trials within 28 days before randomization and used any test drugs or medical devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With a Response of Overall Success(clinical response and microbiological response)[Complicated Urinary Tract Infection (cUTI)] | at Test of Cure (TOC) visit (Day 12-23)
Proportion of Participants Who Died Due to Any Cause[Hospital-acquired Bacterial Pneumonia (HABP), Ventilator-associated Bacterial Pneumonia (VABP) and Bloodstream Infection(BSI) Subjects] | Day 28
Proportion of Participants With a clinical response [Complicated Intra-abdominal Infection (cIAI) Subjects] | at Test of Cure (TOC) visit (Day 10-23

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan Universit, Shanghai, China